CLINICAL TRIAL: NCT04509505
Title: The Effect of Waterpipe Smoking on Periodontal Health Among a Sample of Adult Egyptian Patients. A Hospital Based Cross-sectional Study
Brief Title: Effect of Waterpipe Smoking on Periodontal Health
Status: Completed | Type: Observational
Sponsor: Noha Ayman Ghallab (Other)
Responsible Party: Sponsor-Investigator, Noha Ayman Ghallab, Prof. Dr Noha Ayman Ghallab - Professor of Oral Medicine and Periodontology / Cairo University., Cairo University
Organization: Cairo University (Other)
Other Study IDs: Mariam2020
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Waterpipe Smoking; Periodontal Diseases
MeSH Terms: conditions — Water Pipe Smoking; Periodontal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study is to assess the effect of waterpipe smoking on periodontal health, which will be done using a well constructed validated questionnaire. Then a full periodontal examination and x-ray evaluation will be done for all of the participants.

DETAILED DESCRIPTION:
The primary outcome of the study is to assess the effect of waterpipe smoking on periodontal health, it will be assessed by questions about smoking habits, including smoking mode as well as duration (heads smoked per day) and extent of use (age of initiation and number of sessions per week) of waterpipe smoking.

A full periodontal examination using UNC-15 periodontal probe will be done for all of the participants measuring the CAL, Probing Depth (PD), plaque index (PI), bleeding on probing (BOP) and gingival recession depth (GD). In subjects where attachment loss will be clinically detected, radiographic examination will be performed by digital periapical radiograph to detect the amount of bone loss, then staging will be done according to the new classification by the aid of radiographic examination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is between 18-60 years old.
2. Patient consulting in the outpatient clinic.
3. Provide informed consent.

Exclusion Criteria:

1. Individuals with chronic systemic diseases such as diabetes, endocrine and hematological Pathologies.
2. Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.
3. Pregnant women.
4. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
5. Patients with orthodontic appliances.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
periodontal health condition in waterpipe smokers. | through study completion, an average of 1 year.
  will be assessed from questions about smoking habits, including smoking mode as well as duration and extent of use of waterpipe smoking and measuring the CAL for staging the periodontal condition according to the new classification by the aid of radiographic examination.

SECONDARY OUTCOMES:
Impact of sociodemographic factors on periodontal health | through study completion, an average of 1 year.
  Questions regarding sociodemographic information such as educational level, income and marital status will be analyzed.
Impact of oral hygiene behaviour on periodontal health. | through study completion, an average of 1 year.
  Questions regarding oral health behaviors such as toothbrushing frequency, use of auxiliary aids, dental visits and toothbrushing method will be analyzed too.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Ayman Ghallab, MD, Study Director — Professor of Oral medicine and Periodontology, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Natto S, Baljoon M, Bergstrom J. Tobacco smoking and periodontal health in a Saudi Arabian population. J Periodontol. 2005 Nov;76(11):1919-26. doi: 10.1902/jop.2005.76.11.1919. PMID 16274311
- [Result] Alzyoud S, Veeranki SP, Kheirallah KA, Shotar AM, Pbert L. Validation of the Waterpipe Tolerance Questionnaire Among Jordanian School-Going Adolescent Waterpipe Users. Glob J Health Sci. 2015 Jun 25;8(2):198-208. doi: 10.5539/gjhs.v8n2p198. PMID 26383198
- [Result] Al-Alimi A, Halboub E, Al-Sharabi AK, Taiyeb-Ali T, Jaafar N, Al-Hebshi NN. Independent determinants of periodontitis in Yemeni adults: A case-control study. Int J Dent Hyg. 2018 Nov;16(4):503-511. doi: 10.1111/idh.12352. Epub 2018 Jul 2. PMID 29963753